CLINICAL TRIAL: NCT06438081
Title: Comparison Between Propess (Dinoprostone Controlled Release Pessary) and Cook Double-balloon Catheter for Cervical Priming: a Randomized Controlled Trial
Brief Title: Comparison Between Propess and Cook Double-balloon Catheter for Cervical Priming
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-172
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-05

CONDITIONS: Delivery Problem
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Intervention Model Description: The investigators did a pilot study to compare 5 patients using Cook double-catheter balloon priming and 5 patients using Propess. The investigators found the mean priming to delivery interval was 1971.6 minutes in Propess group and 1212.0 minutes in Cook double-catheter balloon group. The investigators assumed ratio of sample size in Propess and Cook double-catheter balloon was 1:1. In order to achieve 35% reduction of priming to delivery interval, a sample size of 28 is required for Type I error of 0.05, and Type II error of 0.2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cook double-balloon catheter (Active Comparator): Participant is placed in lithotomy position, then to clean vulval and vaginal area, followed by inserting vaginal speculum. Cook double-balloon catheter will be inserted under standard technique. Doctor or midwife guide the cervical ripening balloon with stylet to pass through the cervix. Uterine balloon should be place above level of internal os, then to remove the stylet before further advancing the catheter. Cook double-balloon catheter is further advancing through the cervix until both balloons entered cervical canal. Uterine and vaginal balloons are both inflated with up to 80ml normal saline according to manufacturer recommendation. Maximal duration of balloon placement will be 12 hours. If cervix remains unfavorable after Cook double-catheter balloons, she will be given another Cook double-catheter balloons priming the next day. If cervix remains unfavourable after two balloon priming, elective Caesarean section will be advised.
  Interventions: Combination Product: Cook double-balloon catheter
- Propess (Placebo Comparator): Participant will be firstly confirmed reactive tracing and without regular contraction by non-stress test for 20mins. Propess will be checked its integrity and applied with lubricating jelly before insertion. Propess is inserted to the posterior vaginal fornix. Woman should inform medical staff if they have leaking sensation. After insertion, woman will be advised to lie down and perform non-stress test for 2 hours. Propess will be removed after 24 hours post insertion. Cervical assessment is performed the next day after removal of Propess. Patient with favourable cervix, i.e. Bishop score >= 7, will start artificial rupture of membrane and syntocinon infusion. Patient with unfavorable cervix, i.e. Bishop score <7 is arranged another day of priming by PGE2. If the cervix remains unfavorable after 2 days of pharmacological priming, women will be given a rest day or continued priming by Cook double-balloon catheter.
  Interventions: Combination Product: Cook double-balloon catheter

INTERVENTIONS:
Combination Product: Cook double-balloon catheter — To compare whether Cook double-balloon catheter or Propess able to achieve vaginal delivery with a shorter priming to delivery interval

SUMMARY:
The investigators aimed to compare efficacy and safety of Propess versus Cooks double-balloon catheter for cervical ripening with an unfavorable cervix in term pregnancy.

DETAILED DESCRIPTION:
Previous studies focused on use of PGE2 instead of Propess, which is a preparation of PGE2 packaged in a hydrogel polymer matrix and release 10mg dinoprostone at 0.3mg per hour for 24 hours. Compared with PGE2, Propess can achieve a shorter induction-to-birth interval, a higher rate of vaginal delivery within 24 hours, and a smaller number of vaginal examinations during delivery. However local studies comparing the efficacy and satisfaction of cervical priming between Cook double-balloon catheter and Propess were lacking. The investigators aimed to compare efficacy and safety of Propess versus Cooks double-balloon catheter for cervical ripening with an unfavorable cervix in term pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy
* Cephalic presentation
* Bishop score <7
* At term (>=37+0 weeks of gestation)
* Nulliparous women

Exclusion Criteria:

* Gestation <37weeks
* Multiple pregnancy
* Bishop score <7
* Malpresentation
* Contraindication to vaginal delivery
* Previous Caesarean section
* History of myomectomy
* Maternal fever
* Suspected infection
* Abnormal fetal heart-rate patterns
* Rupture of membranes
* Intrauterine growth restriction
* Not fit for giving consent
* Allergic to Propess or PGE2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Priming to delivery interval | 1 year
  Time for priming (device placement) to delivery interval

SECONDARY OUTCOMES:
Vaginal delivery within 24 hours after priming | 1 year
  delivery within 24 hours
Caesarean section rate | 1 year
  need of resort to Caesarean section and the corresponding indication
Vaginal delivery rate | 1 year
  included instrumental delivery, e.g. vacuum extraction, forcep delivery
Priming to induction interval | 1 year
  Time from priming to induction
Need of induction with oxytocin | 1 year
  Chance of going into spontaneous labor after priming
Amount of oxytocin use | 1 year
  calculate the amount of oxytocin use
Malpresentation after priming | 1 year
  to confirm if cephalic presentation before start of induction
Failed induction rate | 1 year
  defined as cervix failed to dilate to more than 3cm after 12 hours use of oxytocin
Uterine hyperstimulation | 1 year
  defined by a single contraction lasting for more than 2 minutes or more than 5 contractions in 10 minutes for 30 minutes
Suspected intrauterine infection rate | 1 year
  infection rate that require antibiotics treatment
Primary postpartum haemorrhage | 1 year
  Blood loss >500ml within 24 hours of delivery
Length of hospital stay | 1 year
  calculate length of hospital stay after delivery
Maternal satisfaction with the procedure | 1 year
  on a visual analogue scale to rate maternal satisfaction of from 1 to 5, 5 is better, 1 is worse

CONTACTS AND LOCATIONS:
Overall Officials: Yin Fong Leung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No